CLINICAL TRIAL: NCT05453747
Title: Effectiveness of Stabilization Exercise in Youth Basketball Players With Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hazalgenc2
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Basketball Player; Injury, Ankle
Keywords: exercise; basketball player; jump; kinesiophobia
MeSH Terms: conditions — Ankle Injuries; Motor Activity; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Athletes included in the study; They were divided into two groups as those with ankle injury and those without. After the first measurements and evaluations were made, the athletes were given a program that included strength and stabilization exercises. After 8 weeks, the athletes were evaluated for the second time and the effects of the given exercise program on the athletes were examined.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle injury basketball player (Experimental): Athletes included in the study; They were divided into two groups as those with and without ankle injury . The same exercise program was applied to the same group in both groups.
  Interventions: Other: Exercise
- Basketball player (Active Comparator): The same exercise program was applied to the same group in both groups.
  Interventions: Other: Exercise 2

INTERVENTIONS:
Other: Exercise — After evaluating the age groups and physical characteristics of the athletes under the titles of Warm-Up, Core/Balance/Reactive, Speed/Agility/Quickness, Resistance and Cool-Down, the exercise programs that differ for the athlete under these exercise types are listed with the NASM program and shared with the athletes. During the 8-week period between the 2 evaluations, it was applied 2 days a week on the team's fitness days.
  Arms: Ankle injury basketball player
Other: Exercise 2 — After evaluating the age groups and physical characteristics of the athletes under the titles of Warm-Up, Core/Balance/Reactive, Speed/Agility/Quickness, Resistance and Cool-Down, the exercise programs that differ for the athlete under these exercise types are listed with the NASM program and shared with the athletes. During the 8-week period between the 2 evaluations, it was applied 2 days a week on the team's fitness days.
  Arms: Basketball player

SUMMARY:
Ankle injuries are one of the most common sports injuries. Ankle injuries account for 10% to 30% of all injuries and 5% to 20% of all time-wasting injuries. Athletes involved in sports such as football, basketball, and volleyball are particularly at risk for such injuries, largely due to the running and jumping activities involved. Basketball has one of the highest injury rates of any team sport, with 10 injuries in a 1000 hour period.

DETAILED DESCRIPTION:
The ankle is anatomically strong because of the structure of the bones and ligature that make it. Despite this, ankle injuries are the most common type of injury in sports injuries due to the stress and impact of athletes. It is estimated that 25% of the injuries occurred were ankle injuries. Approximately 85% of ankle injuries are lateral ankle sprain.

In basketball, ankle sprain is the most common type of injury. This is because repeated jumps, landings and sudden changes of direction in the nature of basketball. Due to degeneration in the bond structure as a result of ankle sprained, balance problems are also seen in athletes. Therefore, it is important that athletes evaluate the jump performance. In order to better understand the type and severity of injury of athletes, it is necessary to assess not only the physical characteristics but also the anxiety of physical activity and the relationship between this anxiety and injury, as fear of moving in athletes can develop as physical and psychological maturity is not developed enough during the pub period. The fear of moving can negatively affect the healing phases of the injured athlete, or even delay healing.

Plyometric training has been proven to improve muscle strength and power production. In addition, regular exercise can lead to significant improvements in postural control, jumping, sprinting, diversion speed and agility performance in young basketball players. Fear of re-injury is the fear of being vulnerable to painful re-injury even though physical recovery has been achieved. This situation also has an effect on psychological changes such as movements to protect the muscles, insecurity and focusing problems in the physiologically injured area. Studies show that fear of re-injury also influences muscle activation patterns, influencing muscle recovery, neuromuscular function, and rehabilitation outcomes. As a result, this delays the return to sports.

ELIGIBILITY:
Inclusion Criteria:

Between 14-18 years old Become a licensed male basketball player Playing in the Istanbul League of the Turkish Basketball Federation 5 days a week, more than 1.5 hours a day to train

Exclusion Criteria:

Played a match in the 48 hours before the assessment No lower extremity injury other than ankle

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
OptoJump | 8 weeks
  The optojump photoelectric system is a device that is easy to transport and relatively cost-effective. The device is a 96 LED system with a sensor and a transmitter capable of optical measurement. The system can be activated with 2 cameras and at least 2 Optojump bars. The data is recorded via a computer. The system creates a network and it has the ability to detect even 1/1000 seconds of interruption to this network. It can measure data such as time to fall, time to stay in the air, speed, acceleration, number of steps, step length, power, step time. In our study, the data obtained by making the athletes squat jump with Optojump were recorded.
The Tampa Kinesiophobia Scale | 8 weeks
  LThis scale includes questions about fear of movement and is a frequently used scale in musculoskeletal injuries and is a question-answer scale consisting of 17 questions used in sports-related injuries over orthopedic injuries. The questions cover the variables of injury, re-injury, fear and avoidance of movement in the person's work or job-related movements. Likert scale consisting of 1, 2, 3 and 4 points (1: I strongly disagree, 4: I strongly agree) is used in the TSK. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia. It is recommended to use the total score in studies.

SECONDARY OUTCOMES:
Y Balance Test | 8 weeks
  Y Balance Test is a simple but reliable test used to evaluate dynamic balance. Y balance test; It is a dynamic test performed in a one-leg stance that requires strength, flexibility, and proprioception and was developed by Plisky et al. It features a central rectangular base plate 2.54 cm above the ground and 1.5 m long strips in each of the 3 directions. The athlete stands on the soleplate and reaches for each strip with his foot. The score is recorded as the point at which the indicator block was pushed closest to the stance leg.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided